CLINICAL TRIAL: NCT01744366
Title: An Open-label, Multi-centre, Randomised, Parallel-group Trial, Comparing Efficacy and Safety of Degarelix One-month Dosing Regimen With Goserelin in Chinese Patients With Prostate Cancer Requiring Androgen Ablation Therapy
Brief Title: One Month Degarelix/Comparator Treatment for Prostate Cancer in Chinese Population
Acronym: PANDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000006
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Degarelix (Experimental): Degarelix 240/80 mg
  Interventions: Drug: Degarelix
- Goserelin (Active Comparator): Goserelin 3.6 mg
  Interventions: Drug: Goserelin

INTERVENTIONS:
Drug: Degarelix
  Arms: Degarelix
Drug: Goserelin
  Arms: Goserelin

SUMMARY:
One month degarelix/comparator treatment for prostate cancer in Chinese population

ELIGIBILITY:
Inclusion Criteria:

* Chinese male over 18 years
* Adenocarcinoma of the prostate
* Relevant disease status based on lab values and as judged by the physician
* Life expectancy of at least a year

Exclusion Criteria:

* Previous hormonal treatment for prostate cancer
* Considered to be candidate for curative therapy
* Risk or history of any serious or significant health condition
* Has received an investigational drug within the last 28 days and no previous treatment with degarelix

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Cumulative probability of testosterone at castrate level (≤0.5 ng/mL) | Day 28 to Day 364

SECONDARY OUTCOMES:
Proportion of patients with testosterone levels ≤0.5 ng/mL | at Day 3
Percentage change in prostate-specific antigen (PSA) | from baseline to Day 28
Changes in testosterone and PSA levels | Day 0 to 364
Significant changes in laboratory values | Day 0 to Day 364
Significant changes in vital signs | Day 0 to Day 364
Significant changes in body weight | Day 0 to Day 364
Frequency and severity of adverse events | Day 0 to Day 364
Cumulative probability of no PSA failure | Day 0 to Day 364
  PSA failure defined as two consecutive (at least two weeks apart) increase of 50 percentage and at least 5ng/mL increase compared to nadir

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (29):
- China (29):
  - Cancer Institute & Hospital. Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Affiliated Southwest Hospital of 3rd Military Medical University of People's Liberation Army, Chongqing, Chongqing Municipality
  - 1st Afilliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - 2nd.Affiliated Hospital of Xi'an Jiaotong University College of Medicine, Xi’an, Shanxi
  - 1st Hospital Affiliated to Zhejiang University Medical School, Hangzhou, Zhejiang
  - Beijing Hospital of Ministry of Health, Beijing
  - Peking Union Hospital, Beijing
  - Peking University 3rd Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - 1st Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Hunan Province People's Hospital, Changsha
  - People's Hospital of Sichuan, Chengdu
  - 2nd Hospital Affiliated to Zhejiang University Medical School, Hangzhou
  - 1st Hospital of Lanzhou University, Lanzhou
  - 1st Affiliated Hospital of Nanchang University, Nanchang
  - 1st Affiliated Hospital of Nanjing Medical University, Nanjing
  - Drum Tower Hospital Affiliated to Nanjing University Medical School, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Huashan Hospital of Fudan University, Shanghai
  - Shanghai 5th People's Hospital affilicated to Fudan University, Shanghai
  - Shanghai Changhai Hospital, Shanghai
  - 1st Hospital Affiliated to China Medical University, Shenyang
  - 2nd Hospital Affiliated to Suzhou University, Suzhou
  - 2nd Hospital of Tianjin Medical University, Tianjin
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - 1st People's Hospital of Wuxi, Wuxi

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976